CLINICAL TRIAL: NCT01221415
Title: A Comparison of Ultrasound and Nerve Stimulator Techniques for Nerve Localization in Regional Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: not enough manpower
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Leslie Thomas, Anesthesiologist, Ochsner Health System
Other Study IDs: 2007.127.A; 2007.127.A (Other: Ochnser Clinic Foundation Institutional Review Board)
Record Dates: First submitted 2010-07-21; First posted 2010-10-15 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Orthopedic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Interscalene Ultrasound: Subjects having orthopedic surgery requiring an interscalene peripheral nerve block and randomized to have the ultrasound used to locate the nerve.
- Interscalene Nerve Stimulator: Subjects having orthopedic surgery requiring an interscalene peripheral nerve block and randomized to have the nerve stimulator used to locate the nerve.
- Popliteal Ultrasound: Subjects having orthopedic surgery requiring an popliteal peripheral nerve block and randomized to have the ultrasound used to locate the nerve.
- Popliteal Nerve Stimulator: Subjects having orthopedic surgery requiring an popliteal peripheral nerve block and randomized to have the nerve stimulator used to locate the nerve.
- Femoral Ultrasound: Subjects having orthopedic surgery requiring an femoral peripheral nerve block and randomized to have the ultrasound used to locate the nerve.
- Femoral Nerve Stimulator: Subjects having orthopedic surgery requiring an femoral peripheral nerve block and randomized to have the nerve stimulator used to locate the nerve.

SUMMARY:
The primary objective of this study is to compare ultrasound versus nerve stimulator techniques for nerve localization when performing peripheral nerve blocks. Specifically the investigators will be performing Popliteal, Femoral, and Interscalene nerve blocks. The investigators will be looking for differences in 1) time taken to locate the target nerve and inject local anesthetic 2) time from injection of local anesthetic to adequate surgical anesthesia 3) effectiveness of block 4) incidence of vascular puncture 5) incidence of adverse events 6) patient satisfaction.

DETAILED DESCRIPTION:
After obtaining informed consent, subjects will be randomized to either the ultrasound or nerve stimulator groups as the method for nerve localization prior to peripheral block placement.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical status I-III
* Arthroscopic knee surgery or Lower leg/foot surgery as well as shoulder arthroscopy
* Outpatient status
* Patient preference for a regional anesthetic
* Subjects should be capable of giving informed consent

Exclusion Criteria:

* Allergy to:

  * Local anesthetics
  * Hydromorphone
  * Propofol
  * Midazolam
* Patient refusal
* Infection at the injection site
* Peripheral Neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older undergoing outpatient knee arthroscopy or lower leg/foot surgery as well as shoulder arthroscopy.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
time from injection of local anesthetic to adequate surgical anesthesia | within the first 45 minutes after injection of local anesthestic

SECONDARY OUTCOMES:
effectiveness of block | within 1 hour of injection
time taken to locate the target nerve and inject local anesthetic | within 45 minutes prior to injection
incidence of vascular puncture | within 30 minutes of injection
incidence of adverse events | within 2 weeks of the day of surgery
patient satisfaction | within 2 weeks of the date of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Thomas, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Result] Domingo-Triado V, Selfa S, Martinez F, Sanchez-Contreras D, Reche M, Tecles J, Crespo MT, Palanca JM, Moro B. Ultrasound guidance for lateral midfemoral sciatic nerve block: a prospective, comparative, randomized study. Anesth Analg. 2007 May;104(5):1270-4, tables of contents. doi: 10.1213/01.ane.0000221469.24319.49. PMID 17456685
- [Result] Marhofer P, Schrogendorfer K, Wallner T, Koinig H, Mayer N, Kapral S. Ultrasonographic guidance reduces the amount of local anesthetic for 3-in-1 blocks. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):584-8. doi: 10.1016/s1098-7339(98)90086-4. PMID 9840855